CLINICAL TRIAL: NCT04730349
Title: Phase 1/2 Study of Bempegaldesleukin in Combination With Nivolumab in Children, Adolescents, and Young Adults With Recurrent or Refractory Malignancies (PIVOT IO 020)
Brief Title: A Study of Bempegaldesleukin (BEMPEG: NKTR-214) in Combination With Nivolumab in Children, Adolescents and Young Adults With Recurrent or Treatment-resistant Cancer
Acronym: PIVOT IO 020
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Business objectives have changed
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Nektar Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CA045-020; 2020-000854-85 (EudraCT Number)
Record Dates: First submitted 2021-01-26; First posted 2021-01-29 (Actual); Results first posted 2023-03-24 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Ependymoma; Ewing Sarcoma; High-grade Glioma; Leukemia and Lymphoma; Medulloblastoma; Miscellaneous Brain Tumors; Miscellaneous Solid Tumors; Neuroblastoma; Relapsed, Refractory Malignant Neoplasms; Rhabdomyosarcoma
Keywords: B-cell leukemia/lymphoma/non-Hodgkin lymphoma (NHL); BEMPEG; Bempegaldesleukin; CD122-Biased Agonist; CD122-Biased Cytokine; Check point inhibitor; Ependymoma; Ewing sarcoma; High-grade glioma (HGG)/diffuse intrinsic pontine glioma (DIPG); Immunotherapy; IL-2; IL-2 Receptor Agonist; Leukemia and lymphoma; Medulloblastoma; Melanoma; Miscellaneous brain tumors; Miscellaneous solid tumors; Neuroblastoma; Nivolumab; NKTR-214; NIVO; Non-rhabdomyosarcoma soft-tissue sarcomas; Opdivo®; Pediatric cancer; Pediatric malignancy; Rhabdomyosarcoma
MeSH Terms: conditions — Ependymoma; Sarcoma, Ewing; Glioma; Leukemia; Lymphoma; Medulloblastoma; Neuroblastoma; Recurrence; Neoplasms; Rhabdomyosarcoma; Leukemia, B-Cell; Lymphoma, Non-Hodgkin; Melanoma | interventions — Nivolumab; bempegaldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- A1W Dosing schema (Experimental)
  Interventions: Biological: Nivolumab; Biological: NKTR-214
- A1F Dosing schema (Experimental)
  Interventions: Biological: Nivolumab; Biological: NKTR-214
- A2W Dosing schema (Experimental)
  Interventions: Biological: Nivolumab; Biological: NKTR-214
- A2F Dosing schema (Experimental)
  Interventions: Biological: Nivolumab; Biological: NKTR-214
- Part B: Cohort B1 Neuroblastoma (Experimental)
  Interventions: Biological: Nivolumab; Biological: NKTR-214
- Part B: Cohort B2 Ewing sarcoma (Experimental)
  Interventions: Biological: Nivolumab; Biological: NKTR-214
- Part B: Cohort B3 Rhabdomyosarcoma (Experimental)
  Interventions: Biological: Nivolumab; Biological: NKTR-214
- Part B: Cohort B4 Miscellaneous solid tumors (Experimental)
  Interventions: Biological: Nivolumab; Biological: NKTR-214
- Part B: Cohort B5 NHL/leukemia (Experimental)
  Interventions: Biological: Nivolumab; Biological: NKTR-214
- Part B: Cohort B6 High-grade glioma (Experimental)
  Interventions: Biological: Nivolumab; Biological: NKTR-214
- Part B: Cohort B7 Medulloblastoma and Embryonal Tumors (Experimental)
  Interventions: Biological: Nivolumab; Biological: NKTR-214
- Part B: Cohort B8 Ependymoma (Experimental)
  Interventions: Biological: Nivolumab; Biological: NKTR-214
- Part B: Cohort B9 Miscellaneous brain tumors (Experimental)
  Interventions: Biological: Nivolumab; Biological: NKTR-214

INTERVENTIONS:
Biological: Nivolumab — Specified dose on specified days
  Other Names: BMS-936558-01
Biological: NKTR-214 — Specified dose on specified days
  Other Names: Bempegaldesleukin (BEMPEG)

SUMMARY:
The purpose of this study is to first, in Part A, assess the safety, tolerability and drug levels of Bempegaldesleukin (BEMPEG) in combination with nivolumab and then, in Part B, to estimate the preliminary efficacy in children, adolescents and young adults with recurrent or treatment-resistant cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age < 18 years for Part A and Part B
* Age up to 30 years for Part B Cohorts B2, B3 and B4
* Must have received standard of care therapy and there must be no potentially curative treatment available
* Histologically confirmed with malignant neoplasms that are refractory, relapsed, or curative treatments are lacking
* Must have measurable or evaluable disease based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 for solid tumors, Response Assessment in Neuro-Oncology (RANO) or Response Assessment in Pediatric Neuro-Oncology (RAPNO) for central nervous system tumors, International Pediatric Non-Hodgkin Lymphoma Response Criteria for non-Hodgkin lymphoma (NHL), revised International Neuroblastoma Response Criteria (INRC) for neuroblastoma, modified National Comprehensive Cancer Network (NCCN) Criteria for acute lymphoblastic leukemia, and modified Cheson et al International Working Group criteria for acute myeloid leukemia
* Lansky play score for age ≤ 16 years or Karnofsky performance score for age > 16 years assessed within 2 weeks of enrollment must be ≥ 60

Exclusion Criteria:

* Osteosarcoma, T-cell/Natural Killer (NK) cell leukemia/lymphoma, and Hodgkin's lymphoma
* Need for > 2 antihypertensive medications for management of hypertension (including diuretics)
* Known cardiovascular history, including unstable or deteriorating cardiac disease, within the previous 12 months prior to screening
* Inadequately treated adrenal insufficiency
* Active, known, or suspected autoimmune disease
* Active infection requiring systemic therapy within 14 days prior to first dose
* Condition requiring systemic treatment with either corticosteroids or other immunosuppressive medications within 14 days of start of study treatment
* Prior allogeneic stem cell transplant
* Previous severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection either suspected or confirmed within 4 weeks prior to screening

Other protocol-defined inclusion/exclusion criteria apply

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (18):
- United States (2):
  - Local Institution - 0029, Little Rock, Arkansas
  - Local Institution - 0011, St Louis, Missouri
- Australia (4):
  - Local Institution - 0001, Randwick, New South Wales
  - Local Institution, South Brisbane, Queensland
  - Local Institution - 0002, Parkville, Victoria
  - Local Institution - 0003, Perth, Western Australia
- France (4):
  - Local Institution - 0013, Villejuif, Val-de-Marne
  - Local Institution - 0014, Lyon
  - Local Institution - 0016, Marseille
  - Local Institution - 0015, Paris
- Germany (3):
  - Local Institution - 0038, Hamburg
  - Local Institution - 0039, Tübingen
  - Local Institution - 0037, Würzburg
- Local Institution - 0027, Milan, Italy
- Spain (4):
  - Local Institution - 0009, Madrid, Madrid, Comunidad de
  - Local Institution - 0008, Barcelona
  - Local Institution - 0059, Seville
  - Local Institution - 0028, Valencia

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 15 participants were treated in Part A. Study did not progress to Part B; therefore, no participants enrolled in Part B.
Groups:
- Part A: Bempegaldesleukin (0.006 mg/kg)+ Nivolumab (4.5 mg/kg): Bempegaldesleukin 0.006 mg/kg + Nivolumab 4.5 mg/kg administered intravenously every 3 weeks
- Part A: Bempegaldesleukin (0.006 mg/kg)+ Nivolumab (360 mg): Bempegaldesleukin 0.006 mg/kg + Nivolumab 360 mg administered intravenously every 3 weeks
Period: Overall Study
Arm/Group | Part A: Bempegaldesleukin (0.006 mg/kg)+ Nivolumab (4.5 mg/kg) | Part A: Bempegaldesleukin (0.006 mg/kg)+ Nivolumab (360 mg)
Started (Started = Started treatment) | 8 | 7
Completed (Completed = Completed treatment) | 1 | 2
Not Completed | 7 | 5
Not completed — Participant withdrew consent | 1 | 0
Not completed — Disease progression | 6 | 4
Not completed — Study drug toxicity | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Bempegaldesleukin (0.006 mg/kg)+ Nivolumab (4.5 mg/kg) | Part A: Bempegaldesleukin (0.006 mg/kg)+ Nivolumab (360 mg) | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Continuous [Mean (Standard Deviation); unit: Years] | 7.5 (3.9) | 14.9 (1.5) | 10.9 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 4 | 6 | 10
  Unknown or Not Reported | 3 | 1 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race
  Participants
    White | 6 | 5 | 11
    Black or African American | 1 | 0 | 1
    Other | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLTs) - Part A
Description: Number of participants with dose-limiting toxicities (DLTs). DLTs were collected and evaluated for Part A within the DLT evaluation period, which started on Cycle 1 Day 1 (first dose) and ended at Day 42 (42 days after first dose of the study therapy).
Time Frame: From first dose to 42 days after first dose
Population: All treated participants in Part A
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Bempegaldesleukin (0.006 mg/kg)+ Nivolumab (4.5 mg/kg) | Part A: Bempegaldesleukin (0.006 mg/kg)+ Nivolumab (360 mg)
Number analyzed (Participants) | 8 | 7
Participants | 0 | 0

2. Primary Outcome: Number of Participants With Adverse Events (AEs) - Part A
Description: Number of participants with adverse events (AEs). An AE is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Time Frame: From first dose to 30 days after last dose (up to approximately 6 months)
Population: All treated participants in Part A
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Bempegaldesleukin (0.006 mg/kg)+ Nivolumab (4.5 mg/kg) | Part A: Bempegaldesleukin (0.006 mg/kg)+ Nivolumab (360 mg)
Number analyzed (Participants) | 8 | 7
Participants | 8 | 7

3. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) - Part A
Description: Number of participants with serious adverse events (SAEs). SAE is defined as any untoward medical occurrence that, at any dose results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is an important medical event.
Time Frame: From first dose to 30 days after last dose (up to approximately 6 months)
Population: All treated participants in Part A
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Bempegaldesleukin (0.006 mg/kg)+ Nivolumab (4.5 mg/kg) | Part A: Bempegaldesleukin (0.006 mg/kg)+ Nivolumab (360 mg)
Number analyzed (Participants) | 8 | 7
Participants | 6 | 5

4. Primary Outcome: Number of Participants With Drug-Related Adverse Events - Part A
Description: Number of participants with drug-related adverse events. An AE is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Time Frame: From first dose to 30 days after last dose (up to approximately 6 months)
Population: All treated participants in Part A
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Bempegaldesleukin (0.006 mg/kg)+ Nivolumab (4.5 mg/kg) | Part A: Bempegaldesleukin (0.006 mg/kg)+ Nivolumab (360 mg)
Number analyzed (Participants) | 8 | 7
Participants | 6 | 6

5. Primary Outcome: Number of Participants With Adverse Events Leading to Discontinuation - Part A
Description: Number of participants with adverse events leading to discontinuation. An AE is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Time Frame: From first dose to 30 days after last dose (up to approximately 6 months)
Population: All treated participants in Part A
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Bempegaldesleukin (0.006 mg/kg)+ Nivolumab (4.5 mg/kg) | Part A: Bempegaldesleukin (0.006 mg/kg)+ Nivolumab (360 mg)
Number analyzed (Participants) | 8 | 7
Participants | 2 | 3

6. Primary Outcome: Number of Participants Who Died - Part A
Description: Number of participants who died.
Time Frame: From first dose to 30 days after last dose (up to approximately 6 months)
Population: All treated participants in Part A
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Bempegaldesleukin (0.006 mg/kg)+ Nivolumab (4.5 mg/kg) | Part A: Bempegaldesleukin (0.006 mg/kg)+ Nivolumab (360 mg)
Number analyzed (Participants) | 8 | 7
Participants | 2 | 0

7. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) - Part A
Description: Pharmacokinetics (PK) of bempegaldesleukin and nivolumab derived from serum concentration versus time data.
Time Frame: From first dose to 30 days after last dose (up to approximately 6 months)
Population: Data was not and will never be collected
Arm/Group | Part A: Bempegaldesleukin (0.006 mg/kg)+ Nivolumab (4.5 mg/kg) | Part A: Bempegaldesleukin (0.006 mg/kg)+ Nivolumab (360 mg)
Number analyzed (Participants) | 0 | 0

8. Primary Outcome: Trough Observed Concentration (Ctrough) - Part A
Description: Pharmacokinetics (PK) of bempegaldesleukin and nivolumab derived from serum concentration versus time data.
Time Frame: From first dose to 30 days after last dose (up to approximately 6 months)
Population: Data was not and will never be collected
Arm/Group | Part A: Bempegaldesleukin (0.006 mg/kg)+ Nivolumab (4.5 mg/kg) | Part A: Bempegaldesleukin (0.006 mg/kg)+ Nivolumab (360 mg)
Number analyzed (Participants) | 0 | 0

9. Primary Outcome: Area Under the Plasma Concentration (AUC) - Part A
Description: Pharmacokinetics (PK) of bempegaldesleukin and nivolumab derived from serum concentration versus time data.
Time Frame: From first dose to 30 days after last dose (up to approximately 6 months)
Population: Data was not and will never be collected
Arm/Group | Part A: Bempegaldesleukin (0.006 mg/kg)+ Nivolumab (4.5 mg/kg) | Part A: Bempegaldesleukin (0.006 mg/kg)+ Nivolumab (360 mg)
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Participants were assessed for all-cause mortality from their first dose until study completion (up to approximately 13 months). SAEs and Other AEs were assessed from first dose to 150 days after last dose of study therapy (up to approximately 11 months).
Arm/Group | Part A: Bempegaldesleukin (0.006 mg/kg)+ Nivolumab (4.5 mg/kg) | Part A: Bempegaldesleukin (0.006 mg/kg)+ Nivolumab (360 mg)
All-Cause Mortality (participants affected / at risk) | 7/8 | 2/7
Serious Adverse Events (participants affected / at risk) | 8/8 | 5/7
Other Adverse Events (participants affected / at risk) | 8/8 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Bempegaldesleukin (0.006 mg/kg)+ Nivolumab (4.5 mg/kg) (N=8) | Part A: Bempegaldesleukin (0.006 mg/kg)+ Nivolumab (360 mg) (N=7)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Influenza like illness (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 2
Skin wound (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 2
Brain oedema (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Bempegaldesleukin (0.006 mg/kg)+ Nivolumab (4.5 mg/kg) (N=8) | Part A: Bempegaldesleukin (0.006 mg/kg)+ Nivolumab (360 mg) (N=7)
Anaemia (Blood and lymphatic system disorders) | 1 | 3
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 2
Hypoacusis (Ear and labyrinth disorders) | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 1
Eye pain (Eye disorders) | 0 | 1
Photophobia (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 3
Tooth discolouration (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 2
Asthenia (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Fatigue (General disorders) | 4 | 2
Generalised oedema (General disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 1 | 2
Pyrexia (General disorders) | 2 | 3
COVID-19 (Infections and infestations) | 0 | 1
Conjunctivitis (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 0 | 1
Lymphangitis (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1
Vaginal infection (Infections and infestations) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 3
Aspartate aminotransferase increased (Investigations) | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Lymphocyte count decreased (Investigations) | 1 | 3
Neutrophil count decreased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ataxia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 2
Dysgeusia (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 2
Neuralgia (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Behaviour disorder (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Sleep disorder (Psychiatric disorders) | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Scrotal oedema (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 3 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
On 14-Apr-2022, a joint decision was made to end the clinical development program for bempegaldesleukin in combination with nivolumab, resulting in the termination of this study. This results disclosure report provides analyses from CA045-020 Part A safety analyses only. Part B of the study (expansion phase) did not enroll any participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-28): https://cdn.clinicaltrials.gov/large-docs/49/NCT04730349/Prot_SAP_000.pdf